CLINICAL TRIAL: NCT01758666
Title: A Clinical Research on the Relation of Blood Drug Concentration and Calcium Folinate Rescued in High-dose MTX Therapy
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIH-WAC-201205001
Record Dates: First submitted 2012-08-30; First posted 2013-01-01 (Estimated); Last update posted 2015-12-22 (Estimated); Status verified 2012-12

CONDITIONS: Osteosarcoma
MeSH Terms: conditions — Osteosarcoma | interventions — Methotrexate; Leucovorin

ARMS (1):
- Methotrexate and Calcium folinate (Experimental)
  Interventions: Drug: Methotrexate,Calcium folinate

INTERVENTIONS:
Drug: Methotrexate,Calcium folinate

SUMMARY:
At present, the most effective drugs to osteosarcoma include ADM,DDP,,HD-MTX,IFO and so on.The effective rate of single drug was about 30%, and if the chemotherapy contains HD-MTX, the survival rate can reach about 60%, so the HD-MTX is the most important component in patients of osteosarcoma.

Studies have shown that, MTX efficacy and adverse reactions were associated with blood concentration level and duration, selecting the right time and dose to give CF is the critical point.

ELIGIBILITY:
Inclusion Criteria:

1. Proved by pathology in 60 cases of osteosarcoma patients
2. PS ≤ 2, survival period is more than 6 months
3. Normal function of liver and kidney
4. No chemotherapy contraindication, patients treat with high dose methotrexate
5. Get signed written informed consent form
6. Have a good compliance with take blood and follow-up

Exclusion Criteria:

Ages: 12 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 40 (Estimated)
Dates: Start 2012-09; Primary Completion 2016-11 (Estimated); Study Completion 2016-12 (Estimated)

PRIMARY OUTCOMES:
blood concentration of MTX | up to 3 years

SECONDARY OUTCOMES:
other adverse reaction | up to 3 years

CONTACTS AND LOCATIONS:
Overall Officials: Chen Wang, Study Chair — Tianjin Medical University Cancer Institute and Hospital